CLINICAL TRIAL: NCT07321496
Title: The Most Demanding Match Periods: Should GPS Data be Normalized for Performance and Fatigue Monitoring in Soccer?
Brief Title: The Most Demanding Match Periods: Should GPS Data be Normalized
Status: Active, not recruiting | Type: Observational
Sponsor: University of Maia (Other)
Responsible Party: Principal Investigator, Filipe Silvano Pinto Maia, Principal Investigator, University of Maia
Other Study IDs: MDP_01
Record Dates: First submitted 2025-12-20; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Most Demanding Periods; Sport
Keywords: soccer; intensity; training load

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Soccer Players: Soccer players enrolled in the research project
  Interventions: Other: Assessment of most demanding periods in soccer

INTERVENTIONS:
Other: Assessment of most demanding periods in soccer — The most demanding periods will be compared over 3 different time windows: 1, 3 and 5 minutes. Both High speed running and sprint distances will be observed.

SUMMARY:
To date, the characterization of Most Demanding Periods (MDPs) in soccer has relied almost exclusively on absolute metrics, suggesting that the peak demands currently reported in the scientific literature are inherently shaped by these fixed thresholds. This reliance on such absolute metrics may lead to an under- or overestimation of the true relative intensity experienced by each player, thus limiting the accuracy of MDPs interpretation. Therefore, exploring whether normalized thresholds alter the magnitude of MDPs across a range of time windows (1, 3 and 5 minutes) is crucial to better understand how the most demanding passages of match play manifest when player-specific capacities are considered. Consequently, the aim of the present study was to compare the MDPs derived from absolute and normalized thresholds for HSR and sprinting.

ELIGIBILITY:
Inclusion Criteria:

* Soccer players competing at the highest national level

Exclusion Criteria:

* Injured athletes

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: Male Soccer players competing at the highest national level, free from injuries during the period of data analysis.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Distance covered | 1 minute, 3 minute, 5 minute

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade da Maia, Maia, Portugal

IPD SHARING:
Plan to Share IPD: Undecided